CLINICAL TRIAL: NCT06896162
Title: PROGRESS: Precision Oncology Using Genomic Reflexive Evaluations for Study Selection and Survival
Acronym: PROGRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2437-DCT
Record Dates: First submitted 2025-03-14; First posted 2025-03-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor Malignancies; Metastatic Cancer; Breast Cancer; Colorectal Cancer; Lung Cancer; Bladder Cancer
Keywords: next-generation sequencing (NGS); expert review of NGS; precision oncology; precision oncology navigator; genome informed therapy (GIT); biomarker-directed clinical trials
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: hybrid decentralized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The potential candidates for genome-informed targeted therapy (Other): Potential candidates have a stage IV solid tumor malignancy (breast, lung, colorectal, and bladder cancer) for whom NGS testing is planned to be obtained before first or second-line therapy.
  Interventions: Other: Expert Review; Other: Blood or tissue samples collection.; Other: The Precision Oncology Navigation

INTERVENTIONS:
Other: Expert Review — Expert reflexive review of next-generation sequencing (NGS) results will be visible in electronic health records (EPIC) for provider review at the University of North Carolina Health System. Expert review will include recommendations for Genome-informed therapy (GIT), identification of available clinical trials, recommendations for additional testing, and/or referrals for genetic counseling.
Other: Blood or tissue samples collection. — Blood or tissue samples will be collected for next-generation sequencing (NGS) per standard of care.
Other: The Precision Oncology Navigation — The precision oncology navigator will coordinate the collection of blood and /or tissue for next-generation sequencing (NGS), as well as order the NGS if not already ordered. Precision oncology navigator will also assist in NGS financial aid applications, if applicable.

SUMMARY:
This is a hybrid decentralized, single-arm, interventional study designed to evaluate the impact of precision medicine navigation and reflexive expert review of next-generation sequencing (NGS) for patients with stage IV solid tumor malignancies (breast, lung, colorectal, and bladder cancers).

The purpose of this study is to investigate whether intervention from a centralized precision oncology navigator and expert review of NGS results by the precision oncology pharmacist will increase ordering of Level 1/2 genome informed therapy (GIT) compared to an estimated historical rate of 15%. Secondary endpoints will assess the impact of a centralized precision oncology navigator and expert review of NGS results on enrollment in biomarker-directed clinical trials and overall survival at 2 years after return of NGS results. The study will take approximately 12 months for enrolment and 2 years of follow-up after the date of NGS results.

DETAILED DESCRIPTION:
Despite data supporting a survival benefit in many cancers, rates of NGS testing and subsequent GIT are reported to be low in real-world data sets. Rates of multigene panel-based testing and targeted therapy use are reported to be higher at NCI-designated cancer centers compared to other practice types, even when they are associated with a "hub" site. Molecular tumor boards have demonstrated improvements in overall survival in lung cancer, but these models rely on consults being placed by treating physicians and/or significant institutional resources. Many studies evaluating interventions to increase the use of genome informed therapy (GIT) focus on a single cancer type, thereby hindering the ability to operationalize supportive interventions broadly across all cancer types. Given the collective body of data supporting meaningful clinical improvements when patients have access to GIT, we want to study if interventions that make NGS test ordering and interpretation easier for clinicians will increase the rate of orders for GIT. The use of a centralized precision oncology navigator to facilitate completion of NGS testing, expert clinical review from a clinical pharmacist, and documented clinical decision support embedded in the electronic health record represents a unique and more easily scalable model than full molecular tumor board reviews.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria

* Written informed consent was obtained to participate in the study and HIPAA authorization for release of personal health information.
* Subjects are willing and able to comply with study procedures based on the judgment of the investigator.
* Age ≥ 18 years at the time of consent.
* ECOG or Karnofsky Performance Status of 0-2.
* Documented Stage IV solid tumor malignancy: NSCLC, CRC, Breast or Bladder Cancer
* The treating provider deems Next Generation Sequencing (NGS) testing appropriate and plans to consider results in either first- or second-line therapy in the metastatic setting
* A genomic tumor test has not been ordered or has been ordered but not resulted.

Exclusion Criteria:

• Subjects with an active concurrent malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The rate of genome informed therapy (GIT) orders | 2 years
  The rate of genome informed therapy (GIT) orders for Level 1/2 GIT will be compared against an estimated baseline historical GIT order.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival of enrolled patients who receive precision oncology navigation order facilitation and reflexive expert review of their Next Generation Sequencing (NGS) result reporting to the date of death for any cause.
The rate of genome informed therapy (GIT) orders by site | 2 years
  The rate of orders for Level 1/2 genome informed therapy (GIT) at each site.
The rates of consent to UNC Health biomarker-selective clinical trials | 2 years
  The rates of consent to the University of North Carolina (UNC) Health biomarker-selective clinical trial will be calculated. A subgroup analysis of rates of consent by site may be performed.
The reasons for non-consent | 2 years
  Among enrolled patients, if a biomarker-selective clinical trial is identified on expert review of Next Generation Sequencing (NGS) results, reasons for non-consent will be collected.
Overall Survival in subjects who are eligible for Level 1/2 genome-informed therapy (GIT) | 2 years
  To determine the overall survival (OS) after the return of Next Generation Sequencing (NGS) results in those deemed eligible for Level 1/2 genome-informed therapy (GIT) in patients who receive precision oncology navigator order facilitation and reflexive expert review of results.
The rates of referrals for full Molecular Tumor Board | 2 years
  The rates of referrals for full Molecular Tumor Board review in patients who receive precision oncology navigator order facilitation and reflexive expert review of results will be calculated.
The combined rate of orders for Level 1/2 GIT and consent to biomarker-directed clinical trials | 2 years
  To determine the combined rate of orders for Level 1/2 genome-informed therapy (GIT) and consent to biomarker-directed clinical trials open at UNC. Health site in patients who receive precision oncology navigator order facilitation and reflexive expert review of results.
The time between the date of NGS results and the Level 1/2 GIT order date | 2 years
  The time between the date of Next Generation Sequencing (NGS) results and the order date of Level 1/2 GIT will be calculated for those with GIT orders and reported by the site. The median time will be reported for enrolled patients.
Reasons for lack of Level 1/2 GIT orders in eligible subjects | 2 years
  Reasons why patients deemed eligible for Level 1/2 genome-informed therapy (GIT) by expert review do not have orders for GIT will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Lee, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials